CLINICAL TRIAL: NCT03574857
Title: Prospective Comparison of Metolazone Versus Chlorothiazide for Acute Decompensated Heart Failure With Diuretic Resistance
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Emily Burns, Principle Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20455
Record Dates: First submitted 2018-04-16; First posted 2018-07-02 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure Acute; Cardiovascular Diseases
Keywords: Loop diuretics; Heart failure; Diuretic resistance; Thiazide diuretics
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases | interventions — Metolazone; Chlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metolazone (Active Comparator): Metolazone 5 mg by mouth once daily for 2 days
  Interventions: Drug: Metolazone Oral Tablet
- Chlorothiazide (Active Comparator): Chlorothiazide 500 mg IV once daily for 2 days
  Interventions: Drug: Chlorothiazide Injection

INTERVENTIONS:
Drug: Metolazone Oral Tablet — Day 1: Metolazone 5 mg PO Day 2: Metolazone 5 mg PO
  Other Names: Zaroxolyn
  Arms: Metolazone
Drug: Chlorothiazide Injection — Day 1: Chlorothiazide 500 mg IV Day 2: Chlorothiazide 500 mg IV
  Other Names: Diuril
  Arms: Chlorothiazide

SUMMARY:
The primary objective of the study is to compare efficacy of metolazone and chlorothiazide as add-on therapy in patients refractory to loop diuretics with heart failure with a reduced ejection fraction (HFrEF). This will be a single-center randomized pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Admitted for acute decompensated HF with left ventricular ejection fraction (LVEF) <40%
* Refractory fluid overload:
* Unresponsive (<500 mL net negative over previous 24 hours) AND ineffective diuresis (determined by HF team) to moderate intensity push or low intensity continuous infusion loop diuretic (80 mg IV furosemide or equivalent bumetanide dose of 4 mg)
* English or Spanish-speaking subjects
* Willing and able to comply with study procedures

Exclusion Criteria:

* Baseline thiazide use prior to admission or prior to study enrollment
* Renal replacement therapies (RRT) or glomerular filtration rate (GFR) <30 mL/min at the time of enrollment
* Pregnant women
* Cognitive impairment
* Prisoners
* Left ventricular assist devices (LVAD) or temporary mechanical circulatory support devices
* History of cardiac transplant
* Reported allergy to thiazides
* No enteral access or unable to take medications enterally
* Palliative diuretics
* Systolic blood pressure (SBP) <90 mm Hg prior to randomization
* Patients receiving concomitant lithium therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Net urine output at 24 hours | 24 hours
  Milliliters of urine output minus the oral plus intravenous intake

SECONDARY OUTCOMES:
Net urine output at 48 hours | 48 hours
  Milliliters of urine output minus the oral plus IV intake
Net fluid balance over 12 hours | 24 hours
  the net fluid balance over 12 and 24 hours prior to the addition of metolazone or chlorothiazide compared to the 12 hours after addition of the study drug
Net fluid balance over 24 hours | 48 hours
  Net fluid balance over 24 hours prior to the addition of metolazone or chlorothiazide compared to the 24 hours after addition of the study drug
Weight change | 48 hours
  Change in documented weight in kg at 48 hours after starting metolazone or chlorothiazide

OTHER OUTCOMES:
Electrolyte disturbances | 48 hours
  Frequency of hypokalemia, hypomagnesemia, hyponatremia
Worsening renal function | 48 hours
  increase in serum creatinine greater that 0.5 mg/dL from the patient's baseline value on the day of the first dose of chlorothiazide or metolazone
Hospital length of stay | Assessed until hospital discharge, an average of 7 days
  Number of days hospitalized
ICU length of stay | Assessed until hospital discharge, an average of 7 days
  Number of days patient is located in an ICU
In-hospital mortality | Assessed until hospital discharge, an average of 7 days
  Incidence of in-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States